CLINICAL TRIAL: NCT06701981
Title: Etude De L'Effet De Filtres Sur L'Eblouissement D'Inconfort
Brief Title: Study on the Effect of Filters on Discomfort Glare on Healthy Adults
Acronym: PREVIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WS10399; 2024-A00934-43 (Registry Identifier: ANSM RCB)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Glare
Keywords: glare; filter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glare discomfort measures with filters (Experimental)
  Interventions: Other: Filter comparison

INTERVENTIONS:
Other: Filter comparison — Three filters will be compared on light discomfort thresholds using the Lumiz 100™ device

SUMMARY:
The goal of this clinical trial is to evaluate the glare protection provided by two filters compared to no filter. Using the Lumiz 100™ device (a headset with gradually increasing light), participants will measure their discomfort thresholds under three different conditions (one per filter). Each measurement will be repeated three times. The study requires a single visit of 2 hours for each participant. Glare protection will be quantified by comparing discomfort thresholds across the no-filter condition and the two studied filters.

ELIGIBILITY:
Inclusion Criteria:

* A willing person, fluent in French, inclined to follow protocol, capable of reading and understanding the information form, and able to give their free and informed consent.
* Beneficiary of the French Social Security system
* Aged 18 to 65 years
* No or moderate ocular correction (Spherical prescription for distance vision: in the range [-8.00 to +6.00 D]* (negative cylinder) for each eye; Cylindrical prescription for distance vision: in the range [0 to -4.00 D] for each eye; Anisometropia ≤ 2.00 D on the equivalent sphere)
* Correct vision with prescription glasses (Corrected visual acuity +0.10 logMAR or better (distance vision / high contrast / photopic luminance)
* Regular user of sunglasses at least in bright light conditions

Exclusion Criteria:

* Age < 18 years (i.e., no minors in accordance with Article L1121-7 of the Public Health Code of "Code de Santé Publique")
* Pregnant, parturient, or breastfeeding women (Article L1121-5 of the Public Health Code of "Code de Santé Publique")
* Persons deprived of liberty by judicial or administrative decision and persons hospitalized without consent under Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8, and persons admitted to a health or social institution for purposes other than research
* Adults incapable or unable to express their consent (Article L1121-8 of the Public Health Code of "Code de Santé Publique")
* Participant in the exclusion period of another biomedical research study
* Participant who cannot be contacted in case of emergency
* All categories of persons particularly protected under French law are excluded from this research (Articles L1121-5 to L1121-9 of the Public Health Code)
* Employees at the Institut des Sciences de la Vision or EssilorLuxottica
* Ocular pathology that may affect vision (e.g., glaucoma involving visual field loss, maculopathy involving visual acuity loss, or retinitis pigmentosa causing significant discomfort in poorly or overly lit environments)
* Neurological deficit, including a history of epileptic pathology or regular or severe migraines
* Ocular surgery affecting vision (e.g., refractive surgery, cataract surgery, or iridectomy)
* Ocular or head trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Light discomfort thresholds | 2 hours
  Amount of light (in lux) that produce a defined discomfort level (just perceptible or really disturbing)

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Lacan, Phd, Study Director — Essilor International
Locations (1):
- Institut des Sciences de la Vision, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No